CLINICAL TRIAL: NCT03206827
Title: Effects of Dietary Plant and Animal Proteins on Biomarkers of Colorectal Cancer and Type 2 Diabetes in Healthy Adults
Brief Title: Effect of Plant and Animal Proteins on Biomarkers of Colorectal Cancer and Type 2 Diabetes in Healthy Adults (ScenoProt)
Acronym: ScenoProt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Natural Resources Institute Finland (Other Government); Makery Ltd, Finland (Unknown)
Responsible Party: Principal Investigator, Anne-Maria Pajari, Adjunct Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ScenoProt-HY
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer; Type2 Diabetes
Keywords: colorectal cancer; type 2 diabetes; diet; plant protein; animal protein
MeSH Terms: conditions — Colorectal Neoplasms; Diabetes Mellitus, Type 2 | interventions — Plant Proteins; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 70% animal, 30% plant proteins in diet (Active Comparator): Dietary proteins from animal sources 70% and from plant sources 30%, representing an average Finnish diet consumed at the moment.
  Interventions: Other: 70% animal, 30% plant proteins in diet
- 50% animal, 50% plant proteins in diet (Experimental): Dietary proteins from animal sources 50% and from plant sources 50%, containing at most 500 g red meat/week (according to the current Finnish Nutrition Recommendations).
  Interventions: Other: 50% animal, 50% plant proteins in diet
- 30% animal, 70% plant proteins in diet (Experimental): Dietary proteins from animal sources 30% and from plant sources 70%.
  Interventions: Other: 30% animal, 70% plant proteins in diet

INTERVENTIONS:
Other: 70% animal, 30% plant proteins in diet — Diet contains 70% of proteins from animal sources (beef, pork, chicken, dairy products, fish) and 30% from plant sources (bread and cereals).
  Arms: 70% animal, 30% plant proteins in diet
Other: 50% animal, 50% plant proteins in diet — Diet contains 50% of proteins from animal sources (beef, pork, chicken, dairy products, fish) and 50% from plant sources (bread and cereals, legumes, nuts, seeds, soy products).
  Arms: 50% animal, 50% plant proteins in diet
Other: 30% animal, 70% plant proteins in diet — Diet contains 30% of proteins from animal sources (beef, pork, chicken, dairy products, fish) and 70% from plant sources (bread and cereals, legumes, nuts, seeds, soy products).
  Arms: 30% animal, 70% plant proteins in diet

SUMMARY:
The aim of this study is to investigate the effects of dietary plant and animal proteins on gut metabolism and markers for colorectal cancer as well as blood protein metabolites and markers for type 2 diabetes in healthy adults. The study participants will be stratified into three groups with different protein composition in diets: 1) animal 70%/plant 30%; 2) animal 50%/plant 50% and 3) animal 30%/plant 70%. The participants will get part of their diet as ready foods or raw material to promote their compliance. The participants will also get personal advice for their diets. Blood, stool and urine samples will be collected in the beginning and in the end of the 12 week intervention, as well as phenotype measures like BMI, blood pressure and body composition. The participants will also fill food diary before and in the end of the intervention.

DETAILED DESCRIPTION:
A human intervention study with healthy volunteers will be carried out to compare the effects of animal and plant-based protein sources on gut metabolism and markers for colorectal cancer as well as blood protein metabolites and markers for type 2 diabetes.

The study will be done in parallel-design, randomized fashion, with healthy human volunteers aged 20 - 69 years. Exclusion criteria will be as follows: strict vegan, regular user of fish oil or other food supplements, extreme sports, inflammatory bowel disease, colon irritable, celiac disease, continuous antibiotics or less than three months of the latest antibiotics use, type 2 diabetes and hormonal, liver or kidney disease. Duration of the intervention will be 12 weeks.

Intervention groups will be as follows (n=50/group):

Group 1: Dietary proteins from animal sources 70% and from plant sources 30%, representing an average Finnish diet consumed at the moment.

Group 2: Dietary proteins from animal sources 50% and from plant sources 50%, containing at most 500 g red meat/week (according to the current Finnish Nutrition Recommendations).

Group 3: Dietary proteins from animal sources 30% and from plant sources 70%.

The intake of total protein will be kept at similar level compared to habitual, but intakes of fat and carbohydrates may vary as composing a diet with plant-based protein sources inevitably causes changes for example in dietary fibre intake. We will aim at controlling other potential dietary confounders to the extent that is possible in a whole-diet approach. This will ensure the feasibility of the diets and facilitate future applications in dietary practices at the population level.

Before starting the intervention, the persons will get dietary advice how to fulfill their diets. They will get part of foods free to help to implement the diets and to enhance compliance.

Blood, urine and fecal samples will be collected at the baseline (at the beginning of the intervention) and at the end of the intervention. Dietary intake and food consumption during the intervention will be followed by 3-day food records in the beginning and at the end of the intervention period. Nutrient intakes will be calculated using AIVO program.

The following data collection and analyses will be carried out at the beginning and at the end of intervention:

* height, weight, waist circumference
* body composition by bioelectrical impedance analysis
* resting blood pressure, hemoglobin
* fasting lipid profile in the blood (total cholesterol, LDL and HDL, triglycerides)
* fasting glucose and insulin, HbA1c in the blood
* markers for low-grade inflammation in the blood: hs-CRP, cytokines such as IL-1beta, IL-6, IL-10
* protein metabolomics in the blood
* markers of nutritional status in the bood: vit. D25-OH, carotenoids, vitamin C and B12, alkyl resorcinols
* urea/nitrogen in the urine
* measures of gut metabolism and risk markers for colorectal cancer: total N-nitroso compounds in the feces, plant-derived polyphenol metabolites in the feces, concentration of bile acids, cytotoxicity and genotoxicity assays of fecal water samples in 2D and 3D colon cancer cell cultures and gut microbiota analyses.

ELIGIBILITY:
Inclusion Criteria:

Healthy, no exclusion criteria listed below.

Exclusion Criteria:

Strict vegan, food allergies, oral medication for any allergies, regular use of food supplements, extreme sports, inflammatory bowel disease, colon irritable, caeliac disease, any kind of cancer within 5 years, continuous antibiotics or less than three months of the latest antibiotics use, type 1 or 2 diabetes, hormonal, liver or kidney disease, pregnancy, lactation.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Changes in the composition of gut microbiota and glucose metabolism as measures of modification of dietary protein composition | 12 weeks
  The composition of gut microbiota is measured using HITChip phylogenetic microarray. Glucose tolerance test is carried out to analyze glucose metabolism in the beginning and in the end of the intervention.
Changes in the intake of nutrients and nutritional status of participants as a measure of diet modification | 12 weeks
  The changes in the markers for nutritional status in the blood: vit. D25-OH, carotenoids, vitamin C and B12, ferritin, alkyl resorcinols. The intake of nutrients is calculated from 4-day food diaries.

SECONDARY OUTCOMES:
Changes in the concentrations of metabolites derived from plant and animal-based foods in fecal water and urine | 12 weeks
  Concentrations of metabolites derived from plant-based foods in fecal water are measured using UPLC (ultra performance liquid chromatography). Concentrations of fecal nitroso compounds as a measure of red meat consumption is measured as apparent total nitroso compounds.
Genotoxicity testing of human fecal water in 2D and 3D cell cultures | 12 weeks
  Fecal water is isolated from fecal samples collected in the beginning and in the end of intervention period. The samples are tested for markers of genotoxicity in 2D and 3D cell cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Maria Pajari, PhD, Principal Investigator — University of Helsinki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saarinen M, Pellinen T, Kostensalo J, Nousiainen J, Joensuu K, Itkonen ST, Pajari AM. Dietary climate impact correlates ambiguously with health biomarkers- a randomised controlled trial in healthy Finnish adults. Eur J Nutr. 2025 Feb 18;64(2):95. doi: 10.1007/s00394-025-03609-w. PMID 39964546
- [Derived] Pellinen T, Paivarinta E, Isotalo J, Lehtovirta M, Itkonen ST, Korkalo L, Erkkola M, Pajari AM. Replacing dietary animal-source proteins with plant-source proteins changes dietary intake and status of vitamins and minerals in healthy adults: a 12-week randomized controlled trial. Eur J Nutr. 2022 Apr;61(3):1391-1404. doi: 10.1007/s00394-021-02729-3. Epub 2021 Nov 27. PMID 34837522
- [Derived] Itkonen ST, Paivarinta E, Pellinen T, Viitakangas H, Risteli J, Erkkola M, Lamberg-Allardt C, Pajari AM. Partial Replacement of Animal Proteins with Plant Proteins for 12 Weeks Accelerates Bone Turnover Among Healthy Adults: A Randomized Clinical Trial. J Nutr. 2021 Jan 4;151(1):11-19. doi: 10.1093/jn/nxaa264. PMID 32939557